CLINICAL TRIAL: NCT01945528
Title: Pilot Randomized Controlled Trial to Evaluate Safety and Efficacy of Percutaneous Needle Tenotomy With Platelet Rich Plasma (Leukocyte Depleted)in Epicondylitis
Brief Title: Platelet Rich Plasma (PRP) in Chronic Epicondylitis
Acronym: B-PRPtendon
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jose Ignacio Martin (Other Government)
Responsible Party: Sponsor-Investigator, Jose Ignacio Martin, Jose Ignacio Martin, Basque Health Service
Organization: Basque Health Service (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-000478-32; 2013-000478-32 (EudraCT Number)
Record Dates: First submitted 2013-09-16; First posted 2013-09-18 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Epicondylitis
Keywords: Platelet Rich Plasma; tendinopathy; epicondylitis; ultrasound; injection therapy; needle tenotomy
MeSH Terms: conditions — Tendinopathy | interventions — Lidocaine; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- US-guided tenotomy with PRP (Experimental): ultrasound guided percutaneous tenotomy with PRP injection each alternate week for a total of two interventions
  Interventions: Drug: US-guided tenotomy with PRP
- US-guided tenotomy with lidocaine (Active Comparator): ultrasound-guided percutaneous needle tenotomy with lidocaine injection each alternate week for a total of two interventions
  Interventions: Drug: US-guided tenotomy with lidocaine

INTERVENTIONS:
Drug: US-guided tenotomy with PRP — Blood will be drawn from the patient from the patient's unaffected arm. the anti-coagulated blood will be centrifuged and pure-PRP (without leukocytes) collected.
  Local anesthetic (lidocaine) will be infiltrated into the subcutaneous tissue of the lateral elbow, after which a single skin portal and multiple longitudinal and transversal penetrations of the tendon will be performed; PRP will be delivered in multiple depots during the procedure
  Other Names: pure-PRP (without leukocytes)
  Arms: US-guided tenotomy with PRP
Drug: US-guided tenotomy with lidocaine — Blood will be drawn from the patient from the patient's unaffected arm. Local anesthetic (lidocaine) will be infiltrated into the subcutaneous tissue of the lateral elbow, after which a single skin portal and multiple longitudinal and transversal penetrations of the tendon will be performed; lidocaine will be delivered in multiple depots during the procedure
  Other Names: local anesthetic
  Arms: US-guided tenotomy with lidocaine

SUMMARY:
Background Tendinopathy is a difficult problem to manage and can result in significant patient morbidity. Currently, the clinical use of PRP in painful tendons is widespread but its efficacy remains controversial. Current experimental research postulates different efficiency among PRP formulations.Recent reviews showed that most clinical studies in tendinopathies have been performed with L-PRP. The investigators aim to examine the efficacy of pure-PRP in the management of epicondylitis.

The investigators hypothesized that pure PRP associated to needling intervention can enhance tendon healing in epicondylitis, improve function and reduce pain.

Methods and design Randomized double blind controlled trial, a total of 80 patients will be randomly allocated into one of two groups: PRP or control. Interventions: PRP group, ultrasound (US)guided needling associated to delivery of multiple PRP depots each alternate week for a total of two interventions. Control Group: US-guided needling with lidocaine each alternate week for a total of two interventions. Main outcome measure: Changes in pain and activity levels, as assessed by Disabilities of the Arm, Shoulder and Hand (DASH)outcome measure score, before and six months after intervention.The primary end-point is 25% reduction in DASH. The investigators will compare the percentage of patients, in each group, that achieve a successful treatment defined as a reduction of at least 25% in the DASH score.

Secondary outcome measures:Changes in pain and function as assessed by DASH and changes in pain as assessed by the visual analogue scale (VAS)at the 3, 6 and 12 month follow-up. Changes in sonographic features and neovascularity at 3, 6 and 12 months.

ELIGIBILITY:
Inclusion criteria

* Tendinopathy present in either lateral or medial elbow
* Pain by palpation at the lateral or medial epicondyle of the elbow
* Baseline elbow pain >3/10 during resisted wrist extension
* History of at least two periods of elbow pain lasting more than 10 days
* Symptoms lasting at least 3 months or longer
* Body Mass Index between 20 and 35.
* Commitment to comply with all study procedures
* The patient must give written informed consent

Exclusion Criteria:

* Presence of full tendon tear
* Body mass index> 35
* Systemic autoimmune rheumatologic disease (connective tissue diseases and systemic necrotizing vasculitis)
* Poorly controlled diabetes mellitus (glycosylated hemoglobin above 9%)
* Blood disorders (thrombopathy, thrombocytopenia, anemia with Hb <9)
* Patients receiving immunosuppressive treatments
* Received local steroid injection within 3 months of randomization received nonsteroidal antiinflammatory, opioids or oral corticosteroids within 15 days before inclusion in the study
* Severe heart diseasePatients unable to comply with scheduled visits, for work or spend long periods away from their habitual residence.
* Patients with active cancer or cancer diagnosed in the last five years.
* Analytical Diagnosis Hepatitis B, C or HIV infection.
* Pregnant or lactating.
* People who are taking a drug in clinical investigation or participated in any investigational study clinic (with an authorized or not) within 30 days prior to randomization.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-04; Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
changes in the DASH-E score | six months
  percentage of patients that achieve a successful treatment defined as a reduction of at least 25% in the DASH score compared with baseline

SECONDARY OUTCOMES:
Percentage of patients that achieve a successful treatment | three and twelve months
  successful treatment defined as a reduction of greater than 25% of the DASH-E score
Pain reduction as measured by VAS. | three, six and twelve months
  changes in pain rating on a visual analogue scale (VAS)with respect to baseline
changes in echogenicity and vascularity as assessed by Doppler sonography | three, six and twelve months
frequency, severity, intensity and duration of adverse events | three, six and twelve months

CONTACTS AND LOCATIONS:
Overall Officials: Jose I Martin, MD, Principal Investigator — Cruces University Hospital, Osakidetza, Basque Health Service
Locations (2):
- Spain (2):
  - Cruces University Hospital/BioCruces Health Research Institute, Barakaldo, Bizkaia
  - Cruces University Hospital, Barakaldo, Bizkaia

REFERENCES:
- [Background] Andia I, Sanchez M, Maffulli N. Tendon healing and platelet-rich plasma therapies. Expert Opin Biol Ther. 2010 Oct;10(10):1415-26. doi: 10.1517/14712598.2010.514603. PMID 20718690
- [Derived] Karjalainen TV, Silagy M, O'Bryan E, Johnston RV, Cyril S, Buchbinder R. Autologous blood and platelet-rich plasma injection therapy for lateral elbow pain. Cochrane Database Syst Rev. 2021 Sep 30;9(9):CD010951. doi: 10.1002/14651858.CD010951.pub2. PMID 34590307
- [Derived] Martin JI, Atilano L, Merino J, Gonzalez I, Iglesias G, Areizaga L, Bully P, Grandes G, Andia I. Platelet-rich plasma versus lidocaine as tenotomy adjuvants in people with elbow epicondylopathy: a randomized controlled trial. J Orthop Surg Res. 2019 Apr 23;14(1):109. doi: 10.1186/s13018-019-1153-6. PMID 31014382
- [Derived] Martin JI, Atilano L, Merino J, Gonzalez I, Iglesias G, Areizaga L, Bully P, Grandes G, Andia I. Predictors of Outcome Following Tenotomy in Patients with Recalcitrant Epicondylopathy. PM R. 2019 Sep;11(9):979-988. doi: 10.1002/pmrj.12064. Epub 2019 Mar 19. PMID 30609276
- [Derived] Martin JI, Merino J, Atilano L, Areizaga LM, Gomez-Fernandez MC, Burgos-Alonso N, Andia I. Platelet-rich plasma (PRP) in chronic epicondylitis: study protocol for a randomized controlled trial. Trials. 2013 Dec 1;14:410. doi: 10.1186/1745-6215-14-410. PMID 24289799